CLINICAL TRIAL: NCT00299650
Title: Systematic Early Use of Neuromuscular Blocking Agents in ARDS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Pr PAPAZIAN Laurent, ASSISTANCE PUBLIQUE HOPITAUX DE MARSEILLE
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACURASYS; PHRC 2004
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: ARDS
Keywords: ARDS; mortality; mechanical ventilation; pneumonia; muscle relaxants
MeSH Terms: conditions — Pneumonia; Muscle Hypotonia | interventions — cisatracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Active Comparator)
  Interventions: Drug: cisatracurium; Drug: Cisatracurium besilate

INTERVENTIONS:
Drug: cisatracurium
  Arms: B
Drug: Placebo — physiological serum infusion
  Arms: A
Drug: Cisatracurium besilate — Cisatracurium besilate infusion (900mg/day)
  Arms: B

SUMMARY:
The use of neuromuscular blocking agents (NMBA) in ARDS patients has not been extensively investigated. The aim of the study is to show a reduction of the mortality rate of ARDS patients.

DETAILED DESCRIPTION:
The use of neuromuscular blocking agents (NMBA) in ARDS patients has not been extensively investigated. It has been recently demonstrated that a systematic 48-h infusion of NMBA is associated with a significant improvement in oxygenation as compared with a control group (Gainnier et al., Crit Care Med 2004). Moreover, a trend towards a reduction in the mortality rate has been observed. The aim of the study is to show a reduction of the mortality rate of ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* ARDS with a PaO2 / FiO2 < 150 with a PEEP > 5 since less than 48 hrs
* informed consent

Exclusion Criteria:

* NMBA allergy
* Continuous administration of NMBA for ARDS prior inclusion
* Age < 18 yrs
* SAPS II > 70
* Persistent air leak

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the mortality rate of ARDS patients at d90 | 36 months

SECONDARY OUTCOMES:
Mortality at day 28, day 60, day 180 and ICU mortality, Ventilator-free days and alive at day 28 and day 60, Exposure time to FIO2 > 80% or PEEP > 10 cmH2O during the first 7 days, Sedatives and analgesics requirements during the first 7 days | march 2009
Organ failure-free days and alive at day 28, Incidence of barotrauma, Incidence of critical illness neuromyopathy, Incidence of ventilator-associated pneumonia, Quality of life at day 180 | march 2009

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Papazian, MD, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (20):
- France (20):
  - Réanimation polyvalente, Aix-en-Provence
  - Réanimation Polyvalente, Avignon
  - Hôpital Jean Minjoz - Réanimation médicale, Besançon
  - Hôpital Pellegrin - Réanimation médicale, Bordeaux
  - Réanimation médicale, Brest
  - Réanimation chirurgicale, Clermont-Ferrand
  - Hôpital de la Tronche - Réanimation médicale, Grenoble
  - Hôpital de la croix rousse - Réanimation médicale, Lyon
  - Hôpital Ambroise Paré - Réanimation, Marseille
  - Hôpital Sainte-Marguerite - Réanimation médicale, Marseille
  - Réanimation Polyvalente - Hôpital Sainte-Marguerite, Marseille
  - Hôpital Nord - Réanimation, Marseille
  - Réanimation chirurgicale, Montpellier
  - Réanimation médicale, Nice
  - Réanimation chirurgicale, Nîmes
  - Réanimation Médicale, Nîmes
  - Hôpital Saint-Louis - Réanimation médicale, Paris
  - Hôpital Pontchaillou - Réanimation médicale, Rennes
  - Hôpital Bellevue - Réanimation Médicale, Saint-Etienne
  - Réanimation polyvalente, Toulon

REFERENCES:
- [Derived] Guerin C, Papazian L, Reignier J, Ayzac L, Loundou A, Forel JM; investigators of the Acurasys and Proseva trials. Effect of driving pressure on mortality in ARDS patients during lung protective mechanical ventilation in two randomized controlled trials. Crit Care. 2016 Nov 29;20(1):384. doi: 10.1186/s13054-016-1556-2. PMID 27894328
- [Derived] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245